CLINICAL TRIAL: NCT03254901
Title: Detection of Hepatitis C Infection by Oraquick Test Among Health Care Workers in Assiut Governorate and Treatment Outcome Among True Positive Cases
Brief Title: Detection of Hepatitis C Infection by Oraquick Test Among Health Care Workers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hebe Gaafar, principal investigator, Assiut University
Other Study IDs: HCVAssiut
Record Dates: First submitted 2017-08-17; First posted 2017-08-21 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- health care workers: health care workers in Assiut health directorate, Abutig central hospital, El-Quseya central hospital and Sahil selim central hospital in Assiut governorate .All of them will be screened for hepatitis C infection and interviewed about mode of transmission of infection
  Interventions: Other: Screening test by Oraquick test

INTERVENTIONS:
Other: Screening test by Oraquick test — The OraQuick assay uses an indirect immunoassay method to detect hepatitis C antibodies in oral fluid or blood

SUMMARY:
Viral hepatitis is a global health problem affecting hundred millions of people worldwide and considered the main cause of liver cirrhosis, hepatocellular carcinoma and liver transplantation in developing countries.

DETAILED DESCRIPTION:
Hepatitis C is a chronic disease affecting approximately 130-170 million people worldwide. According to the world health organization, annually, more than 399,000 people die from hepatitis C-related liver diseases and 3-4 million people are infected with hepatitis C virus . Approximately 3% of the world's population is estimated to be infected with hepatitis C virus .

Hepatitis C is found worldwide. World health organization documented that Eastern Mediterranean and European regions are the most affected regions, with the prevalence of 2.3% and 1.5% respectively. Prevalence of hepatitis C virus infection in other world health organization regions varies from 0.5% to 1.0%. There are multiple strains ( genotypes) of the hepatitis C virus and their distribution varies by region.

Available data indicate that infection with hepatitis C virus infection varies considerably by country and region and countries believed to have the highest rate of chronic hepatitis C virus infection are Egypt (15 %), Pakistan (4.8 %), and China (3.2 %). However, the true incidence of the disease is not well known in many countries, because acute infection is generally asymptomatic.

The Egyptian Demographic Health Survey ( 2008), which was conducted on a large nationally representative sample, estimated the prevalence of hepatitis C virus antibodies and hepatitis C virus nucleic acid, among the 15-59 years age group, to be 14.7 and 9.8% respectively. On the other hand, the prevalence of hepatitis C virus antibodies and hepatitis C virus nucleic acid, among the 15-59 years age group, to be 10 and 7 % respectively according to the Egyptian Health Issues Survey ( 2015).There was an overall significant reduction of 32 %and 29% in the prevalence of Hepatitis C virus antibody and Hepatitis C virus nucleic acid-positive individuals, respectively, between the Egyptian Demographic Health Survey in 2008 and the the Egyptian Health Issues Survey in 2015.

Hepatitis C virus is a bloodborne virus. It is most commonly transmitted through injecting drug use through the sharing of injection equipment; the reuse or inadequate sterilization of medical equipment, especially syringes and needles in healthcare settings; and the transfusion of unscreened blood and blood products.

hepatitis C virus can also be transmitted sexually and can be passed from an infected mother to her baby; however these modes of transmission are much less common, while it is not spread through breast milk, food, water or by casual contact such as hugging, kissing and sharing food or drinks with an infected person.

ELIGIBILITY:
Inclusion Criteria:

* no inclusion criteria as we select all health care workers at Assiut health directorate. By systematic random sample, every second person from lists of health care workers in Abutig central hospital, El-Quseya central hospital, Sahil selim central hospital will be selected

Exclusion Criteria:

* no exclusion criteria

Ages: 21 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: health care workers in Abutig central hospital, El-Quseya central hospital, Sahil selim central hospital and Assiut health directorate
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
percentage of hepatitis C virus infection among health care workers | six months
  hepatitis C infection is screened by oraquick test the confirmed by hepatitis C nucleic acid testing

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kandeel A, Genedy M, El-Refai S, Funk AL, Fontanet A, Talaat M. The prevalence of hepatitis C virus infection in Egypt 2015: implications for future policy on prevention and treatment. Liver Int. 2017 Jan;37(1):45-53. doi: 10.1111/liv.13186. Epub 2016 Jun 30. PMID 27275625
- [Result] Guidelines for the Screening, Care and Treatment of Persons with Hepatitis C Infection. Geneva: World Health Organization; 2014 Apr. Available from http://www.ncbi.nlm.nih.gov/books/NBK263483/ PMID 25535634
- [Result] Martin NK, Vickerman P, Miners A, Foster GR, Hutchinson SJ, Goldberg DJ, Hickman M. Cost-effectiveness of hepatitis C virus antiviral treatment for injection drug user populations. Hepatology. 2012 Jan;55(1):49-57. doi: 10.1002/hep.24656. Epub 2011 Dec 6. PMID 21898506
- [Result] Lee SR, Yearwood GD, Guillon GB, Kurtz LA, Fischl M, Friel T, Berne CA, Kardos KW. Evaluation of a rapid, point-of-care test device for the diagnosis of hepatitis C infection. J Clin Virol. 2010 May;48(1):15-7. doi: 10.1016/j.jcv.2010.02.018. Epub 2010 Apr 1. PMID 20362493